CLINICAL TRIAL: NCT03116139
Title: 1 R01 HL132358: The Contribution of Contrast Media Exposure to Acute Kidney Injury in Patients Evaluated for Pulmonary Embolism in the Emergency Care Setting: a Prospective, Randomized Trial
Brief Title: Acute Kidney Injury in Patients Undergoing Contrast Exposure: VQ vs. CT
Acronym: VQ/CT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study funding ended prior to planned study accrual and prior to planned completion of all enrolled subjects.
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alice Mitchell, Assistant Professor of Emergency Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VQ/CT; 1R01HL132358-01A1 (NIH)
Record Dates: First submitted 2017-04-03; First posted 2017-04-14 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Acute Kidney Injury; Pulmonary Embolism; Contrast-induced Nephropathy
Keywords: Computed tomography scan; Ventilation-perfusion lung scan; Acute kidney injury; Pulmonary embolism; Contrast-induced nephropathy
MeSH Terms: conditions — Acute Kidney Injury; Pulmonary Embolism | interventions — Ventilation-Perfusion Scan; Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low risk for kidney injury with use of CT (No Intervention): No randomization due to low risk for kidney injury. 100 patients undergoing CTPA with an estimated risk of CIN <10% (CINRisk Score <2)
- Randomized to V/Q (Active Comparator): 300 patients with > 25% estimated risk of CIN (CINRisk Score ≥ 2), randomized to VQ imaging (unexposed control)
  Interventions: Diagnostic Test: V/Q imaging
- Randomized to CT (Active Comparator): 300 patients with > 25% estimated risk of CIN (CINRisk Score ≥ 2), randomized to CT (exposure to iodinated contrast media)
  Interventions: Diagnostic Test: Computed tomography scan

INTERVENTIONS:
Diagnostic Test: V/Q imaging — Standard of care
  Other Names: Ventilation perfusion scan
  Arms: Randomized to V/Q
Diagnostic Test: Computed tomography scan — Standard of care
  Other Names: CT; CTPA
  Arms: Randomized to CT

SUMMARY:
Both, CT scans and VQ scans, are used by doctors to look for pulmonary embolism. The most common reason to order a VQ scan is to avoid the IV dye. The IV dye used for CT scans can cause kidney problems in some patients, called contrast-induced nephropathy or "CIN." This is a kidney problem that usually does not make patients feel any differently or change how they urinate. Most of the time, it can only be found by testing blood several days later. This kind of kidney problem can be very mild and some patients will never have any symptoms, rarely these problems can be severe. Some patients can also have similar kidney problems for many other reasons (reactions to medications, blood pressure problems, etc.) and can even happen in patients that do not get IV dye. That is why doctors are not sure exactly who will have these problems or if using a test that does not use IV dye can prevent this kidney problem. The VQ scan uses a different medication through the IV that is not IV dye and has not been linked to kidney problems. The purpose of this study is to learn if using the test that does not use IV dye (the "VQ scan") instead of a CT scan in some patients can help to prevent kidney problems.

DETAILED DESCRIPTION:
Before the study begins, research personnel will do the following to be sure that patients can be in the study:

* research personnel will talk to the treating physician.
* research personnel will review the patient medical records, blood and urine tests already done for as usual medical care, and chest X-ray.
* research personnel will ask the patients some questions about their health.
* If it has not already been done for usual medical care, patients will be asked to give a urine sample to test for medical conditions that may result in a higher risk of having kidney problems such as having glucose (sugar) in the urine.

If the patient is eligible to continue in the study, the following will also happen at the initial day of enrollment:

* research personnel may draw about 4 tablespoons of blood from the vein or, if from the IV that was (or will be) placed for usual medical care.
* If one of the 100 patients who are at low risk of kidney problems, they will have a CT scan of the chest that was ordered by the doctor.
* Otherwise, the potential subject will be randomly assigned to have either a CT scan of the chest, which will include dye given in an IV, or a VQ scan, that does not use IV dye. One half will have the CT scan and one half will have the VQ scan.
* Potential subjects will also have an ultrasound (a painless sound wave test of the legs to look for a clot in the legs that can cause a clot in the lungs), if the doctor thinks that one is needed, or if the VQ scan is "indeterminate." Indeterminate means that the radiologist, the doctor reading the VQ scan, cannot tell if there is a pulmonary embolism (a clot in your lung). Research personnel expect that less than 5% (5 out of 100) patients will have a VQ scan that is indeterminate. Some patients who have a VQ scan that is indeterminate, may also need to have a CT scan of their chest to be sure that they do or do not have a clot in their lungs.
* research personnel will also save blood and urine samples. Later, these samples will be used to test for electrolytes (salts) and proteins (that may help better predict who will get kidney problems. Subjects will not have to pay for these tests because they will not be used for usual medical care. To protect privacy, research personnel will use a code instead of name to label samples. For this reason, research personnel will not be able to tell the results of these tests.
* If you are not found to be eligible for this study, the reason will be discussed with you and your treating provider. If you are eligible to continue in the study, the following will happen later:
* Subjects will be given an appointment to return to the hospital between 2 and 7 days from the initial visit. As a reminder, research personnel will give subjects a reminder card; research personnel will call and/or text the subjects, and/or email with reminders. If subjects are still in the hospital during this time, research personnel will visit the subjects in the hospital.
* At this appointment research personnel will ask some questions about the health, will take about 4 tablespoons of blood and a urine sample. Blood and urine will be used to test for kidney problems. If these tests do show a kidney problems after having IV dye, research personnel will send a letter to notify subjects and the treating physician.
* In 30 days, research personnel will make 3 attempts to call and ask some questions about the subject's health. If research personnel cannot follow up by telephone, they will also try to contact by text, and/or by mail.
* research personnel will also review medical records in 7 days, 30 days, and in 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years
2. CTPA ordered by the treating provider to evaluate PE.
3. Pre-test probability of PE ≤20% (defined using the PE Pretest Consult Score)
4. For Randomization to CTPA or VQ imaging: Pre-imaging CIN risk ≥25% (CINRisk Score ≥2 points) • A lower-risk subset of 100 patients (CINRisk Score <2) will be enrolled and followed. These patients will complete the CTPA as ordered by their provider (not randomized). Data from this lower-risk subset, along with high-risk patients randomized to CTPA will be used will be used to validate the CINRisk Score, alone and in combination with NGAL and eGFRCYS (Study Aims 1 and 3).

Exclusion Criteria:

1. History of pulmonary surgery or pulmonary infiltrate, mass or effusion on chest radiograph.
2. Clinical instability preventing randomization to CTPA or VQ imaging.
3. Pregnancy or ≤48 hours post-partum
4. Subject unavailability for reasonable follow-up including biological sample collection, serum creatinine measurement, and interview, such as an insecure residence, planned travel or absence, personal or professional obligations, incarceration, and/or other reason preventing follow-up, identified at enrollment.
5. Active renal replacement therapy (hemodialysis or peritoneal dialysis) within 30-days of enrollment or previous physician-directed plans to initiate dialysis within 30-days of the index visit.
6. Prior renal transplant or planned within 30-days of enrollment.
7. Intravascular contrast administration within 14 days prior to enrollment or planned within 7 days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Incidence of AKI at 7 days | 7 days post enrollment
  Percentage of participants with a creatinine increase ≥ 0.3 mg/dL or 1.5 times baseline

SECONDARY OUTCOMES:
Validate the acute kidney injury score, alone and in combination with acute-phase markers of renal dysfunction. | Enrollment
  Compare the incidence of short, mid- and long-term AKI and subsequent health outcomes in patients exposed to iodinated contrast media and unexposed controls.
Validate the acute kidney injury score, alone and in combination with acute-phase markers of renal dysfunction. | 2-7 days post enrollment
  Compare the incidence of short, mid- and long-term AKI and subsequent health outcomes in patients exposed to iodinated contrast media and unexposed controls.
Incidence of AKI at 30 days | 30 days post enrollment
  Percentage of participants with a creatinine increase ≥ 0.3 mg/dL or 1.5 times baseline
Incidence of AKI at 1 year | 1 year post enrollment
  Percentage of participants with a creatinine increase ≥ 0.3 mg/dL or 1.5 times baseline
Incidence of subsequent health outcomes at 30 days in participants who developed AKI | 30 days post enrollment
  Percentage of participants who developed AKI and subsequent health outcomes
Incidence of subsequent health outcomes at 30 days in participants who did not developed AKI | 30 days post enrollment
  Percentage of participants who did not develop AKI, however, did develop subsequent health outcomes
Incidence of subsequent health outcomes at 1 year in participants who developed AKI | 1 year post enrollment
  Percentage of participants who developed AKI and subsequent health outcomes
Incidence of subsequent health outcomes at 1 year in participants who did not developed AKI | 1 year post enrollment
  Percentage of participants who did not develop AKI, however, did develop subsequent health outcomes
Incidence of VTE at 30 days | 30 days post enrollment
  Percentage of participants who developed VTE
Incidence of VTE at 1 year | 1 year post enrollment
  Percentage of participants who developed VTE
Incidence of subsequent health outcomes at 30 days in participants who developed VTE | 30 days post enrollment
  Percentage of participants who developed VTE and subsequent health outcomes
Incidence of subsequent health outcomes at 30 days in participants who did not develop VTE | 30 days post enrollment
  Percentage of participants who did not develop VTE, however, did develop subsequent health outcomes
Incidence of subsequent health outcomes at 1 year in participants who developed VTE | 1 year post enrollment
  Percentage of participants who developed VTE and subsequent health outcomes
Incidence of subsequent health outcomes at 1 year in participants who did not develop | 1 year post enrollment
  Percentage of participants who did not develop VTE, however, did develop subsequent health outcomes
Incidence AKI associated with an elevated AKI risk score | 7 days post enrollment
  Percentage of participants with AKI risk score is >=2
Incidence AKI associated with an elevated AKI risk score or acute phase biomarker | 7 days post enrollment
  Percentage of participants with AKI risk score is >=2 or an abnormal acute phase biomarker
Incidence AKI associated with a non-elevated AKI risk score | 7 days post enrollment
  Percentage of participants with AKI risk score is <2
Incidence AKI associated with a non-elevated AKI risk score and normal acute phase biomarker | 7 days post enrollment
  Percentage of participants with AKI risk score is <2 nor an abnormal acute phase biomarker

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Indiana University Health, Indianapolis, Indiana
  - Corewell Health, Royal Oak, Michigan
  - Baylor, Scott & White Health, Dallas, Texas
  - Intermountain Healthcare, Murray, Utah
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT03116139/Prot_SAP_001.pdf